CLINICAL TRIAL: NCT05870475
Title: A Randomized Controlled Study Evaluating the Efficacy and Safety of Pegylated Interferon α-2b in Combination With Ruxolitinib vs. Pegylated Interferon α-2b Monotherapy for Treating Hydroxyurea-resistant/Intolerant Polycythemia Vera
Brief Title: Pegylated Interferon α-2b in Combination With Ruxolitinib for Treating Hydroxyurea-resistant/Intolerant PV
Acronym: PV
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023018
Record Dates: First submitted 2023-04-10; First posted 2023-05-23 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-05

CONDITIONS: Polycythemia Vera
MeSH Terms: conditions — Polycythemia Vera | interventions — ruxolitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pegylated interferon α-2b in combination with ruxolitinib group (Experimental): Pegylated interferon α-2b in combination with ruxolitinib group: Pegylated interferon α-2b at a starting dose of 180ug, subcutaneous injection once a week; ruxolitinib at a starting dose of 10mg, orally administered twice daily.
  Interventions: Drug: Ruxolitinib; Drug: Pegylated interferon α-2b
- Pegylated interferon α-2b group (Active Comparator): Pegylated interferon α-2b group: Starting dose of 180ug, subcutaneous injection once a week.
  If complete hematological remission is not achieved after 12 weeks of treatment with pegylated interferon α-2b alone, cross-over to the pegylated interferon α-2b plus ruxolitinib group is allowed; if ruxolitinib is not tolerated, cross-over to the pegylated interferon α-2b alone group is allowed.
  Interventions: Drug: Pegylated interferon α-2b

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib at a starting dose of 10mg, orally administered twice daily. If ruxolitinib is not tolerated, cross-over to the pegylated interferon α-2b alone group is allowed.
  Other Names: RUX
  Arms: pegylated interferon α-2b in combination with ruxolitinib group
Drug: Pegylated interferon α-2b — Starting dose of 180ug, subcutaneous injection once a week. If complete hematological remission is not achieved after 12 weeks of treatment with pegylated interferon α-2b alone, cross-over to the pegylated interferon α-2b plus ruxolitinib group is allowed.
  Other Names: PEG IFNα-2b

SUMMARY:
Study purpose: To compare the efficacy and safety of pegylated interferon α-2b in combination with ruxolitinib versus pegylated interferon α-2b alone for treating hydroxyurea-resistant or hydroxyurea-intolerant polycythemia vera.

DETAILED DESCRIPTION:
Study purpose: To compare the efficacy and safety of pegylated interferon α-2b in combination with ruxolitinib versus pegylated interferon α-2b alone for treating hydroxyurea-resistant or hydroxyurea-intolerant polycythemia vera.

The subjects will be randomly divided into two groups:

pegylated interferon alpha-2b combined with ruxolitinib group: pegylated interferon alpha-2b at a starting dose of 180ug will be administered subcutaneously once a week; ruxolitinib at a starting dose of 10mg will be administered orally twice daily.

pegylated interferon alpha-2b group: pegylated interferon alpha-2b at a starting dose of 180ug will be administered subcutaneously once a week.

If complete hematologic remission is not achieved after 12 weeks of treatment with pegylated interferon alpha-2b alone, the subject may be switched to the pegylated interferon alpha-2b combined with ruxolitinib group. If ruxolitinib is not tolerated, the subject may be switched to the pegylated interferon alpha-2b group alone.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old.
* Male or Female.
* Meets the diagnostic criteria for Polycythemia Vera according to WHO-2022.
* Resistant or intolerant to hydroxyurea (based on the 2013 European LeukemiaNet criteria).
* Have not previously received interferon preparations or ruxolitinib treatment, or the washout period between the last use of interferon preparations or ruxolitinib and the first use of the study drug should not be less than 4 weeks.
* Patients with indications for cytoreductive therapy.
* During screening, female hemoglobin (HGB) ≥10g/dL, male hemoglobin (HGB) ≥11g/dL; neutrophil count ≥1.5×109/L; platelet count ≥100×109/L.
* Voluntary written informed consent.

Exclusion Criteria:

* Symptomatic splenomegaly;
* Contraindications to interferon or ruxolitinib therapy;
* Severe or significant comorbidities that may affect the participant's ability to participate in the study, as determined by the investigator;
* History of major organ transplantation;
* Pregnant or breastfeeding women;
* History or current diagnosis of autoimmune thyroid disease (patients with controlled hypothyroidism on oral thyroid hormone replacement therapy may be included);
* Documented evidence of any other autoimmune disease (such as active hepatitis, systemic lupus erythematosus, antiphospholipid antibody syndrome, or autoimmune arthritis);
* Clinically significant bacterial, fungal, mycobacterial, parasitic, or viral infection such as active hepatitis or HIV infection (patients with acute bacterial infections requiring antibiotic treatment should be deferred from screening/enrollment until completion of antibiotic treatment);
* Evidence of severe retinopathy or clinically significant ophthalmologic disease (due to diabetes or hypertension);
* Current clinically significant depression or history of depression, or any suicidal attempt or tendency during screening;
* Active bleeding or thrombotic complications;
* History of any malignant tumor within the past 5 years (except for stage 0 chronic lymphocytic leukemia [CLL], cured basal cell carcinoma, squamous cell carcinoma, and superficial melanoma);
* History of alcohol or substance abuse within the past year;
* Presence of blasts in the peripheral blood within the past 3 months;
* Use of any investigational drug or participation in any other clinical trial within 4 weeks prior to the first dose of the study drug, or failure to recover from any effects of previously administered study drugs;
* The investigator deems the presence of any concurrent condition that may jeopardize the safety of the participant or the compliance to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
The cumulative complete hematologic response (CHR) rate | From the start of study treatment (Week 0) up to the end of Week 24.
  The proportion of patients who can achieve CHR ( defined as hematocrit lower than 45% without phlebotomies; platelet count < 400×109/L, WBC count < 10×109/L for at least 12 weeks) among all patients.

SECONDARY OUTCOMES:
Cumulative CHR rates at Week 36. | From the start of study treatment (Week 0) up to the end of Week 36.
  Cumulative CHR rates at Week 36 will be compared between the two groups.
Cumulative CHR rates at Week 52. | From the start of study treatment (Week 0) up to the end of Week 52.
  Cumulative CHR rates at Week 52 will be compared between the two groups.
Time to CHR | From the start of study treatment (Week 0) up to the end of Week 52.
  The time of reaching CHR will be compared between the two groups.
The CHR rates after crossover | From the start of study treatment (Week 0) up to the end of Week 52.
  The CHR rates within 52 weeks after crossover
The rate of reduction in JAK2V617F, CALR, or MPL gene mutation burden. | From the start of study treatment (Week 0) up to the end of Week 52.
  The rate of reduction in JAK2V617F, CALR, or MPL gene mutation burden will be compared between the two groups.
Impact of therapy on non-driver mutations | From the start of study treatment (Week 0) up to the end of Week 52.
  To compare the proportion of subjects that display change on key non-driver biomarkers of the disease-DNMT3A, ASXL1, TET2 or other mutations.
Change of splenomegaly | From the start of study treatment (Week 0) up to the end of Week 52.]
  All subjects with palpable splenomegaly at baseline will undergo ultrasound examination.
  For subjects with palpable splenomegaly at baseline:
  Improvement - no palpable splenomegaly during clinical treatment visits; No progress - ultrasound examination during clinical treatment visits shows an increase in spleen size of ≤ 25%; Progress - Ultrasound examination during clinical treatment visits shows an increase in spleen size of>25%.
Change of bone marrow pathology | From the start of study treatment (Week 0) up to the end of Week 52
  Bone marrow histological remission defined as the presence of age-adjusted normocellularity and disappearance of trilinear hyperplasia, and absence of grade 1 reticulin fibrosis; no remission defined as the persistence of trilinear hyperplasia; progression defined as disease transformation into post-PV myelofibrosis, myelodysplastic syndrome or acute leukemia.
The incidence of major thrombotic events | From the start of study treatment (Week 0) up to the end of Week 52.
  To compare the incidence of major thrombotic events between the two groups.
The incidence of major bleeding events | From the start of study treatment (Week 0) up to the end of Week 52.
  To compare the incidence of major bleeding events between the two groups.
The incidence of progressing to acute leukemia | From the start of study treatment (Week 0) up to the end of Week 52.
  The incidence of progressing to acute leukemia will be compared between the two groups.
Change in Myeloproliferative Neoplasm Symptom Assessment Form total symptom score | From the start of study treatment (Week 0) up to the end of Week 52.
  To compare the proportion of subjects that display change in Myeloproliferative Neoplasm Symptom Assessment Form total symptom score (0-100 scores, higher scores mean a worse outcome) between different treatment groups.
Change of quality of life using QLQ-C30 V3.0 questionnaire. | From the start of study treatment (Week 0) up to the end of Week 52.
  The QLQ-C30 V3.0 questionnaire consists of 30 questions, with questions 1-28 scoring 1-4 and questions 29 and 30 scoring 1-7. Therefore, this questionnaire has a minimum score of 30 and a maximum score of 126, and the score is directly proportional to the quality of life.
Change of microcirculation disturbance | From the start of study treatment (Week 0) up to the end of Week 52.
  The rate of patients with improvement in microcirculation disturbance (such as pruritus, headache, dizziness, chest tightness, erythematous limb pain and limb paresthesia) will be compared between the two groups
Specific pre-defined toxicity | From the start of study treatment (Week 0) up to the end of Week 52.
  To compare incidence of specific pre-defined toxicity including fatigue, flu-like symptoms, dizziness, injection site necrosis, dyspnea, pain, depression, blurred Vision, insomnia, anorexia, weight Loss, weakness, pruritis, sweating, fever, decreased Libido, hot Flashes, flushing, infection,

OTHER OUTCOMES:
Changes of T lymphocytes | From the start of study treatment (Week 0) up to the end of Week 52.
  Change in the proportion and gene expression profile of T lymphocytes
Changes of B lymphocytes | From the start of study treatment (Week 0) up to the end of Week 52.
  Change in the proportion and gene expression profile of B lymphocytes
Changes of dendritic cells | From the start of study treatment (Week 0) up to the end of Week 52.
  Change in the proportion and gene expression profile of dendritic cells

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China; Rongfeng Fu, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China